CLINICAL TRIAL: NCT05710523
Title: Efficay of Training on Non-pharmacological Therapies With People With Dementia in Nursing Home: Integration Between Learning, Body and Emotions in Synergy (I-ACE). A Randomized Double-blind Controlled Study.
Brief Title: Integration Between Learning, Body and Emotions (I-ACE)
Acronym: I-ACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associazione Ginco Ticino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Burnout, Professional; Dementia; Quality of Life
Keywords: burnout; nursing home staff; dementia; oxytocine; training
MeSH Terms: conditions — Burnout, Professional; Dementia; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The I-ACE training encompasses a training on the non-pharmacological therapies' methodology and a training on awareness of body language which favors a passage from implicit to explicit knowledge. It allows the reading of the subjective relational experience of the care situation by the professional caregiver and a comparison of shared readings of the situation itself by the group of colleagues, and with the residents. Participants will follow:
  Two sessions, each lasting 4 hours, on theoretical introduction to the non-pharmacological therapies' methodology; Ten monthly supervisions, each lasting one and half hours, on discussion of clinical cases and implementation of the non-pharmacological therapies with person with dementia.
  Ten monthly supervisions, each lasting two hours, on theatrical exercises guided by an expert actor, with the help of a psychologist-psychotherapist who promotes understanding and awareness of self-reading in the relationship with the other.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- I-ACE training (Experimental): Participants will receive twenty-two sessions on the non-pharmacological therapies' methodology and on awareness of body language.
  Interventions: Behavioral: I-ACE training
- Standard non-pharmacological therapies (NPT) training (Active Comparator): Participants will receive twelve sessions on the non-pharmacological therapies' methodology.
  Interventions: Other: Standard non-pharmacological therapies (NPT) training
- As usual control group (No Intervention): Participants will continue the usual care activities and non-pharmacological interventions already in use in the Nursing Homes without participating in the training.

INTERVENTIONS:
Behavioral: I-ACE training — The I-ACE training encompasses a training on the non-pharmacological therapies' methodology and a training on awareness of body language which favors a passage from implicit to explicit knowledge. It allows the reading of the subjective relational experience of the care situation by the professional caregiver and a comparison of shared readings of the situation itself by the group of colleagues, and with the residents. Participants will follow:
  Two sessions, each lasting 4 hours, on theoretical introduction to the non-pharmacological therapies' methodology; Ten monthly supervisions, each lasting one and half hours, on discussion of clinical cases and implementation of the non-pharmacological therapies with person with dementia.
  Ten monthly supervisions, each lasting two hours, on theatrical exercises guided by an expert actor, with the help of a psychologist-psychotherapist who promotes understanding and awareness of self-reading in the relationship with the other.
  Arms: I-ACE training
Other: Standard non-pharmacological therapies (NPT) training — The standard NPT training encompasses a training on the non-pharmacological therapies' methodology. Participants will follow:
  Two sessions, each lasting 4 hours, on theoretical introduction to the non-pharmacological therapies' methodology; Ten monthly supervisions, each lasting one and half hours, on discussion of clinical cases and implementation of the non-pharmacological therapies with person with dementia.
  Arms: Standard non-pharmacological therapies (NPT) training

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of training on non-pharmacological therapies (NPT) for people with dementia (PWD) on professional caregivers burnout and well-being in the relationship between caregivers and people with dementia (PWD) living in nursing home.

The main questions it aims to answer are:

* Does I-ACE training, that includes a training in the emotional-behavioral reading of body language and the recognition of one's own emotions and those of others, reduces professional caregiver burnout?
* Does I-ACE training improves the ability to understand and respond to the emotions of the other starting from the signals expressed by the eyes, the activation of the predisposition to the relationship in terms of increase of salivary oxytocin, the sense of competence of the carers, the ethical climate at the workplace and the quality of life of the resident perceived by the team?

Participants will attend twenty-two sessions:

two theoretical meetings on dementia and NPT; ten supervision meetings on the methodology for implementing non-pharmacological therapies based on discussions of cases; ten meetings on the exploration of the bodily aspects involved in the relationship through theatrical exercises. The same cases will be re-discussed in the light of the body-emotional approach.

Researchers will compare the I-ACE group with an active control group and an usual care control group to see if there are improvements in term of professional caregivers burnout, their ability to understand and respond to the emotions of PWD, increase of their levels of salivary oxytocin, sense of competence of the carers, the ethical climate at the workplace and the quality of life of the resident perceived by the team.

DETAILED DESCRIPTION:
The I-ACE study is a complex, single-center, randomized, controlled, single-blind experimental study with three parallel arms: I-ACE training (experimental group), standard NPT training (active control group), and a usual care group. The study aims to evaluate the effectiveness of a year and a half NPT training that includes a theoretical-experiential dimension on the body (I-ACE training), compared to a standard NPT training, and usual care activities. The study involves the professional caregivers of the Nursing Homes of the Canton of Ticino.

Participants in I-ACE study are professional caregivers of 15 Nursing Home in Canton Ticino area. The Nursing Home's responsibles will identify participants responding to inclusion criteria with the help of Principal investigator. The study coordinator (responsible Professor Rita Pezzati) will verify the presence of the inclusion and exclusion criteria. This information will be promptly transferred and kept in an electronic archive protected by a password. Access to the personal computer containing the data will be protected by an access key. In the database, to each subject will be assigned an identification code without references to personal data, which will be kept separately and protected by a keyword known only to the research manager or his delegate. The list of codes relating to the Nursing Homes and the eligible subjects will be delivered to the researcher who will arrange for the randomization. After generating the randomisation sequence, an independent researcher will forward it to the study coordinator for the assignment of the Nursing Homes to each of the three groups, experimental, active control and as usual control (block size (5 x 3 = 15).

In line with similar studies (Gómez-Gascón et al., 2013; Verweij et al., 2018) we have planned three parallel arms with 90 subjects per arm, an estimated medium effect size (d = 0.05), an alpha level of 0.05, and a power of 0.91. Thereafter, a 10% attrition rate due to possible acute clinical conditions interfering with the participation in the study was considered. The power calculation was performed with the programme G*Power 3.1.

ELIGIBILITY:
Inclusion Criteria:

* Length of service more than six months.

Exclusion Criteria:

* Presence of psychiatric illness or other medical condition that prevents participation in the training.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Professional caregivers' burnout | 547 days
  Improvement in professional caregivers' burnout, as measured by the Maslach Burnout Inventory, from pre to post intervention. We expect a significant difference in the experimental group compared with the two control groups.

SECONDARY OUTCOMES:
Professional caregivers' reading the mind in the eyes | 547 days
  Improvement in the ability of professional caregivers to understand and respond to the emotions of the other starting from the signals expressed by the eyes, as measured by the Reading the mind in the eyes test, from pre to post intervention. We expect a significant difference in the experimental group compared to the two control groups.
Salivary oxytocin of professional caregivers | 547 days
  Improvement in the salivary oxytocin of professional caregivers, from pre to post intervention. We expect a significant difference in the experimental group compared to the two control groups.
Professional caregivers' sense of competence | 547 days
  Improvement in the professional caregivers' sense of competence, as measured by the Dementia Care Staff Sense of Competence in Dementia Care Staff Scale, from pre to post intervention. We expect a significant difference in the experimental group compared to the two control groups.
professional caregivers' perception of social capital and ethical climate | 547 days
  Improvement in the professional caregivers' perception of social capital and ethical climate, as measured by the Social capital and ethical climate at the Workplace of a hospital scale (SEW), from pre to post intervention. We expect a significant difference in the experimental group compared to the two control groups.
Quality of life of people with dementia | 547 days
  Improvement in the quality of life of people with dementia perceived from professional caregivers, as measured by the Quality of Life in Late-stage Dementia questionnaire (QUALID), from pre to post intervention. We expect a significant difference in the experimental group compared to the two control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Pezzati, Professor, Principal Investigator — Ginco Ticino Association
Locations (1):
- Nuring Homes of Canton Ticino area, Lugano, Canton Ticino, Switzerland